CLINICAL TRIAL: NCT04392700
Title: A Prospective Randomized Controlled Trial of Tenofovir and Entecavir in the Treatment of Long-term Prognosis in Patients With Hepatitis B-related Hepatocellular Carcinoma After Curative Resection
Brief Title: A RCT of TNF and ENT in the Treatment of Long-term Prognosis With Hepatitis B-related HCC After Curative Resection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhongguo Zhou, professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B2019-05201
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Hepatocellular Carcinoma Recurrent
Keywords: antiviral therapy; hepatocellular carcinoma; prognosis
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Tenofovir; entecavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group A (Experimental): drugs：tenofovir disoproxil fumarate, dose：300mg/d
  Interventions: Drug: Tenofovir disoproxil fumarate 300mg
- group B (Active Comparator): drugs：entecavir dose： 0.5 mg/d
  Interventions: Drug: Entecavir 0.5 mg

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate 300mg — Take the medicine once a day ，300mg/d
  Other Names: Fu Ma Suan Ti Nuo Fu Wei Er Bi Fu Zhi Pian
  Arms: group A
Drug: Entecavir 0.5 mg — Take the medicine once a day，0.5 mg/d
  Other Names: EnTiKaWeiPian(BoLuDing)
  Arms: group B

SUMMARY:
This study evaluates the addition of Tenofovir and Entecavir in the treatment of Hepatitis B-related hepatocellular carcinoma after curative resection in adults. Half of participants will receive Tenofovir disoproxil fumarate, while the other half will receive Entecavir.

DETAILED DESCRIPTION:
Antiviral potency significantly differs among various antiviral agents，Entecavir and tenofovir disoproxil fumarate are equally recommendedas first-line treatments for patients with chronic hepatitis B (CHB). However, it is unclear whether treatment with these drugs is associated with equivalent clinical outcomes,especially impacts the risk of HCC recurrence. Entecavir and tenofovir disoproxil fumarate have comparable efficacy in achieving surrogate end points, including virologic response,but they do by different mechanisms .

Entecavir, a guanosine nucleoside analogue with activity against HBV reverse transcriptase (rt),is efficiently phosphorylated to the active triphosphate form, which has an intracellular half-life of 15 hours. By competing with the natural substrate deoxyguanosine triphosphate, entecavir triphosphate functionally inhibits all three activities of the HBV reverse transcriptase: (1) basepriming, (2) reverse transcription of the negative strand from the pregenomic messenger RNA,and (3) synthesis of the positive strand of HBV DNA.

Tenofovir fumarate is a cyclic nucleoside phosphine diester structural analog of adenosine monophosphate. Tenofovir disoproxil fumarate first needs to be converted to tenofovir by hydrolysis of the diester, followed by phosphorylation of cellular enzymes to form tenofovir diphosphate. Tenofovir diphosphate competes with the natural substrate 5'-deoxyadenosine triphosphate for its involvement in the synthesis of viral DNA, which, after entering the viral DNA strand, can cause DNA elongation to be blocked due to its lack of 3'-OH groups,thereby blocking the replication of the virus. Tenofovir diphosphate is a weak inhibitor of mammalian DNA polymerase alpha, beta and mitochondrial DNA polymerase gamma.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 to 70 years
2. Positive test for hepatitis B surface antigen (HBsAg) and negative tests for antibodies to hepatitis C virus (HCV-Ab) or to human immunodeficiency virus
3. Clinical diagnosis is consistent with HCC and histopathological result of the resected specimens being HCC
4. No previous treatment of HCC and no previous treatment of hepatitis B with nucleoside or nucleotide analogues or both; no previous treatment with interferon or other immunomodulators
5. BCLC stage 0, A or a solitary tumor with a diameter >5cm
6. No extrahepatic metastasisc
7. No radiologic evidence of invasion into major portal/hepatic venous branches
8. Good liver function with Child-Pugh Class A or Child - Pugh Class B (If B Child - Pugh score ≤7 ) and baseline serum alanine aminotransferase (ALT) level less than 3 times the upper limit of normal (reference range <40IU/L), with no history of encephalopathy, ascites refractory to diuretics, esophagogastric variceal bleeding
9. Good renal function (a serum creatinine level<133mmol/L)
10. Negative resection margin (R0 resection)
11. Laboratory blood tests : WBC≥≥3.0×10^9/L ; PLT≥75×10^9/L ; Hb≥100g/L Cr<133mmol/L ; ALT≤ 150U/L ; AST ≤ 120U/L ; ALB≥30g/L ; TBIL≤34mmol/L INR < 1.5 ; APTT < 18 S

Exclusion Criteria:

1. Eligible patients were excluded if they refused to participate
2. Histopathological result of the resected specimens being not HCC
3. History of antiviral therapy
4. History of receive treatment of HCC， include drugs 、radiofrequency ablation transcatheter arterial chemoembolization or resection
5. age﹤ 18 or ﹥70 years
6. Pregnant or lactating women
7. Poor liver function and poor renal function
8. Suffering from other serious acute or chronic physical or mental illness
9. The following occurred before the study began：Myocardial infarction、 Unstable angina、Coronary artery bypass surgery、Cerebrovascular 、 Pulmonary embolism

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 706 (Estimated)
Dates: Start 2019-07-25 (Actual); Primary Completion 2021-07-25 (Estimated); Study Completion 2024-07-25 (Estimated)

PRIMARY OUTCOMES:
Recurrence of HCC | 36 months
  radiologic evidence of tumor recurrence（CT or MRI ） at any time during the following time after liver resection

SECONDARY OUTCOMES:
The number of overall patients | 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China